CLINICAL TRIAL: NCT06380972
Title: A Prospective, Multicenter, Randomized, No-treatmentcontrolled, Evaluator-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of Polycaprolactone Microspherical Injectable to Improve Forehead Contour
Brief Title: A Prospective, Randomized, No-treatment Controlled, Evaluator-blinded Clinical Trial to Evaluate the Efficacy and Safety of Polycaprolactone Microspherical Injectable to Improve Forehead Contour
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AQTIS Medical B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDM6009A-301
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-04

CONDITIONS: Forehead Contouring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the method of endpoint blind evaluation is adopted, that is, it's blinded for the evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polycaprolactone (PCL) Based Facial Injectable (Experimental)
  Interventions: Device: Polycaprolactone (PCL) Based Facial Injectable
- no treatment control (No Intervention)

INTERVENTIONS:
Device: Polycaprolactone (PCL) Based Facial Injectable — Polycaprolactone (PCL) Based Facial Injectable
  Arms: Polycaprolactone (PCL) Based Facial Injectable

SUMMARY:
A Prospective, Multicenter, Randomized, No-treatment-controlled, Evaluator-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of Polycaprolactone Based Facial Injectable to Improve Forehead Contour

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age (whichever is the time of signing informed consent) of either sex;
2. Subjects who are seeking treatment for forehead contour improvement;
3. Subjects with moderate to severe forehead contour deficiency (i.e., ASFS score of 2-3) as evaluated by blinded investigator according to Asian Sloping Forehead Scale (ASFS);
4. Subjects who are in good health and suitable for receiving treatment for forehead contour improvement as assessed by the investigator;
5. Subjects who are willing to sign informed consent, understand and accept the duration of the study, and are able and willing to comply with all requirements, including scheduled treatment, follow-up, and other study procedures (including clinical photography).

Exclusion Criteria:

1. Those with a history of severe allergy or anaphylactic shock or those with a history of allergy which may result in a response to treatment;
2. Those with known allergy to polycaprolactone, carboxymethylcellulose, or any of the ingredients in this product, any local anesthetics such as lidocaine or other amide anesthetics;
3. Those with tattoos, scars, deformities, non-healing wounds, active skin disease or skin inflammation (e.g., herpes, acne, eczema, dermatitis, psoriasis, herpes zoster, etc.), abscess, cancer or pre-cancerous lesions and so forth on the forehead that may affect the evaluation of efficacy or increase the risk of treatment;
4. Those who have received, or plan to receive during the trial, any permanent filler (e.g., polymethyl methacrylate, organic silicon, expanded polytetrafluoroethylene, etc.), autologous fat or unspecified injectables in the frontal region;
5. Those who have received treatment on the forehead such as calcium hydroxyapatite (CaHA), poly-L-lactic acid (PLLA), and polycaprolactone (PCL) within 2 years prior to screening or during the planned trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The response rate for improving the forehead contour is assessed by the blinded investigator using the Asian Sloping Forehead Scale (ASFS) | Month 12

SECONDARY OUTCOMES:
The response rate of forehead contour improvement assessed by blinded investigator using Asian Sloping Forehead Scale (ASFS) | at Months 1, 3, 6 and 9
The response rate of forehead contour improvement assessed by injection investigator using Asian Sloping Forehead Scale (ASFS) | at Months 1, 3, 6, 9 and 12
The global aesthetic improvement rate assessed by the injection investigator based on the Global Aesthetic Improvement Scale (GAIS) | at Months 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Overall Officials: SHENGKANG LUO, Principal Investigator — Guangdong Second People's Hospital
Locations (2):
- China (2):
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isik S, Sahin I. Contour restoration of the forehead by lipofilling: our experience. Aesthetic Plast Surg. 2012 Aug;36(4):761-6. doi: 10.1007/s00266-011-9800-2. Epub 2012 Mar 22. PMID 22434157
- [Background] Hong WJ, Liao ZF, Zeng L, Luo CE, Luo SK. Tomography of the Forehead Arteries and Tailored Filler Injection for Forehead Volumizing and Contouring. Dermatol Surg. 2020 Dec;46(12):1615-1620. doi: 10.1097/DSS.0000000000002561. PMID 32740211